CLINICAL TRIAL: NCT06216938
Title: Phase I Pilot Study of RP1 in Primary Melanoma to Reduce the Risk of Sentinel Lymph Node Metastasis
Brief Title: RP1 in Primary Melanoma to Reduce the Risk of Sentinel Lymph Node Metastasis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yana Najjar (Other)
Collaborators: Replimune Inc. (Industry)
Responsible Party: Sponsor-Investigator, Yana Najjar, Associate Professor of Medicine / Medical oncologist/hematologist, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 22-138
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Melanoma
Keywords: sentinel lymph node (SLN); herpes simplex virus 1 (HSV1); Granulocyte-macrophage colony stimulating factor (GM-CSF)
MeSH Terms: conditions — Melanoma | interventions — MAPRE1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vusolimogene oderparepvec (RP1) (Experimental): Patients will receive 3 doses of RP1 (1.0 mL/injection; 10e6 PFU/mL for the first dose, and 10e7 mL for the subsequent 2 doses). The drug will be injected into the skin at the tumor biopsy site at baseline (day 1), day 15, and day 21, 4-5 weeks prior to SOC WLE and SLNB. Definitive surgery will occur up to 28-35 (± 2 days) days from first injection, to avoid treatment delay.
  Interventions: Biological: Vusolimogene oderparepvec (RP1)

INTERVENTIONS:
Biological: Vusolimogene oderparepvec (RP1) — Vusolimogene Oderparepvec is a genetically modified oncolytic viral strain of the herpes simplex type 1 (HSV-1) virus, with potential oncolytic, immunostimulating and antineoplastic activities.

SUMMARY:
This early-phase study will examine Vusolimogene Oderparepvec, a genetically modified oncolytic viral strain of the herpes simplex type 1 (HSV-1) virus, with potential oncolytic, immunostimulating and antineoplastic activities. Upon administration, vusolimogene oderparepvec specifically targets, infects and replicates in tumor cells and does not infect healthy cells. This results in tumor cell lysis and the release of virus particles which infect and replicate within nearby tumor cells, resulting in tumor cel death. The immune system is activated by the released tumor-associated antigens (TAAs) from the tumor cells creating an anti-tumor immune response against the tumor cells, thereby further killing the tumor cells. The virus itself also elicits a tumor-specific systemic immune and cytotoxic T-lymphocyte (CTL) response, thereby killing nearby non-infected tumor cells.

DETAILED DESCRIPTION:
The majority of the almost 80,000 patients newly diagnosed with melanoma each year in the U.S. present with localized early-stage melanoma (i.e., clinical stage I/II). Per the standard of care (SOC), these patients are treated with a curative intent, including wide local excision (WLE), with additional sentinel lymph node (SLN) biopsy (SLNB) for patients with Breslow ≥ 0.8 mm or < 0.8 mm with ulceration or a positive deep margin. The incidence of SLN metastases significantly increases with the Breslow thickness of the tumor and the presence of ulceration. For T3b (Breslow > 2 mm, with ulceration), the incidence of SLN metastases is 23-42%. For T4b disease (Breslow > 4 mm), this increases up to 63%. As the tumor draining lymph node (TDLN), the SLN is where naïve T cells are first primed. However, this is also the site where melanoma cells initiate tumor mediated immune suppression and form the pre-metastatic niche. Thus, the SLN is a key potential target for local immune therapeutic intervention in early-stage melanoma patients, whereby tumor-mediated immune suppression can be counteracted, and the antitumor immune response can be boosted. As SLN positivity is the single most important prognostic factor in early-stage melanoma, intervention at the SLN may prevent disease recurrence. Almost all patients diagnosed with melanoma will have already undergone a diagnostic biopsy by the time they are seen by medical oncology. The majority undergo shave biopsy by dermatology or their primary care physician, and a smaller proportion have undergone punch or excisional biopsy. Replimune is developing vusolimogene oderparepvec (RP1), an oncolytic immunotherapy. RP1 is a selectively replicating competent herpes simplex virus 1 (HSV-1) that expresses exogenous genes and is administered by intratumoral injection. Local delivery of RP1 following initial biopsy of primary melanoma, prior to SLNB, provides a unique setting to clinically assess the role of the TDLN in the biological efficacy of RP1.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Have a diagnosis of pT3b, T4a or T4b melanoma on biopsy. Patients must have grossly visible residual tumor, or a positive deep or lateral margin on initial biopsy. Patients with uveal melanoma are not eligible.
4. Females of childbearing potential must have a negative beta-human chorionic gonadotropin (β-hCG) test with a minimum sensitivity of 25 IU/L or equivalent units of β-hCG during screening, before the first dose, and a negative urine pregnancy test on days of treatment (Day 1, 15 and 21). For serum and urine pregnancy tests and instructions (see Section 12.2).
5. Female patients of reproductive potential must agree to avoid becoming pregnant and adhere to a highly effective contraception method until 90 days after last dose of RP1 alone. For a definition of highly effective contraceptive methods and instructions of patients and partners (see Section 12.2).
6. Male patients of reproductive potential must agree to avoid impregnating a partner and adhere to a highly effective contraception method until 90 days after last dose of RP1 study agent and refrain from donating sperm during this period. For a definition of highly effective contraceptive methods and instructions of patients and partners (see Section 12.2).

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
7. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
8. Demonstrate adequate organ function. All screening labs should be performed within 30 days of treatment initiation. Baseline labs may be used as screening labs.

Exclusion Criteria:

1. Prior treatment with an oncolytic virus therapy.
2. Has acute or chronic active hepatitis B and C virus infection or known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (HCV) (defined as HCV RNA [qualitative]) or HIV infection.

   Note: No testing for Hepatitis B, Hepatitis C, or HIV is required unless mandated by local health authority or clinically indicated.
3. Had systemic infection requiring IV antibiotics or other serious infection within 14 days prior to dosing.
4. Have active significant herpetic infections or prior complications of HSV-1 infection (e.g., herpetic keratitis or encephalitis).
5. Conditions requiring treatment with immunosuppressive doses (> 10 mg daily prednisone or equivalent) of systemic corticosteroids other than for corticosteroid replacement therapy within 14 days after enrollment. For the definition of replacement therapy (Section 11.0 Supportive Care and Management of Adverse Reactions/Events).
6. Major surgery ≤ 1 week prior to starting study drug. Note: Patients who undergo major surgery must adequately recover prior to starting study treatment.
7. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within four weeks prior to the first dose of study treatment.
8. History of documented allergic reactions or acute hypersensitivity reactions attributed to RP1 or any of its excipients.
9. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacille Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed, however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.

   Note: Available COVID-19 vaccines do not contain live virus.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that will be unfavorable for the administration of study drug or affect the explanation of drug toxicity or AEs or interfere with the patient's participation for the full duration of the study or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
11. Has serious or uncontrolled medical disorders.
12. Has known psychiatric, alcohol abuse, or substance abuse disorders that would interfere with cooperating with the requirements of the study.
13. Is a person deprived of their liberty by a judicial or administrative decision, or an adult person subject to a legal protection measure.
14. Is a solid organ transplant recipient.
15. Has a concurrent malignancy requiring active systemic therapy or ongoing radiation.
16. Patients with tumors that are located near critical structures, such as the carotid artery or portal vein, or scalp lesions presenting with moderate to extensive bone erosion and tumors that may have invaded the heart, great vessels, or other critical structures will not be eligible because these area should not be injected. Injection through an ulcerated area of a lesion should be avoided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Sentinel Lymph Node (SLN) Positivity | Up to 2 years (cohort)
  Proportion of patients with sentinel lymph node lymph node positivity (disease present in lymph node per pathologic assessment).

SECONDARY OUTCOMES:
Incidence of all treatment-emergent adverse events (TEAEs) | Up to 2 years
  Distinct number of patients that experience treatment-emergent adverse events (TEAEs) by highest grade per CTCAE v5.0.
Incidence of ≥ Grade 3 Treatment Emergent Adverse Events (TEAEs) | Up to 2 years
  Distinct number of patients that experience ≥ Grade 3 treatment-emergent adverse events (TEAEs) by highest grade per CTCAE v5.0.
Incidence of Serious Adverse Events (SAEs) | Up to 2 years
  Distinct number of distinct patients that experience Serious Adverse Events (SAEs) by highest grade per CTCAE v5.0.
Incidence of fatal Adverse Events (AEs) | Up to 2 years
  Distinct number of patients that experience fatal Adverse Events (AEs) by highest grade per CTCAE v5.0.
Incidence of all treatment-emergent adverse events (TEAEs) requiring withdrawal from RP1 | Up to 2 years
  Distinct number of patients that experience treatment-emergent adverse events (TEAEs) requiring withdrawal from RP1 by highest grade per CTCAE v5.0.
Recurrence Free Survival (RFS) | Up to 3 years
  Median number of months from start of treatment to recurrence of disease or death from any cause. Recurrence of disease is defined as
Overall Survival (OS) | Up to 3 years
  Median number of months from start of treatment until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yana Najjar, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No